CLINICAL TRIAL: NCT05143333
Title: Cognitive Assessment in COVID Positive Patients Using the DANA App
Brief Title: Cognitive Assessment in COVID-19 Positive Patients Using the DANA App
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: AnthroTronix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00271687
Record Dates: First submitted 2021-12-01; First posted 2021-12-03 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
Keywords: COVID-19 cognition
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post acute COVID-19: Severity of COVID-19 will be determined based on patient classification within the PACT (Johns Hopkins Post-acute COVID-19 Team) clinic. Specifically, patients followed in the PACT-ICU clinic required ICU stays of ≥48 hours and high-flow nasal cannula/non-invasive ventilation or mechanical ventilation. Those followed in the PACT-Base clinic have less severe disease that does not necessitate ≥48 hours in the ICU but does qualify for PACT clinic referral based on either (1) ongoing pulmonary and/or rehabilitation needs at the time of hospital discharge, or (2) persistent pulmonary or functional deficits at 4-6 weeks post infection without hospitalization.
  Interventions: Other: DANA app

INTERVENTIONS:
Other: DANA app — The Defense Automated Neurobehavioral Assessment (DANA) is a battery of cognitive tests delivered via an electronic tablet or smartphone. The platform allows higher temporal precision and frequency of measurement than traditional neuropsychological methods while including previously standardized cognitive tests and allowing individuals to repeatedly self-administer the battery in their own homes without examiner supervision. Hence, the DANA battery bypasses several of the major limitations associated with in-person cognitive exams.

SUMMARY:
The Defense Automated Neurobehavioral Assessment (DANA) is a battery of cognitive tests delivered via an electronic tablet or smartphone. The overarching goal of this study is to evaluate the post-acute trajectory of cognitive functioning in patients hospitalized for COVID-19 using the DANA.

DETAILED DESCRIPTION:
The sequelae of COVID-19 are increasingly appreciated to be systemic and persistent among certain populations. Retrospective review of severe COVID-19 cases revealed increased altered mental status, encephalitis, psychosis, and neurocognitive abnormalities in the three weeks following discharge. During severe COVID-19 infection, there is additional evidence of cerebrovascular events, including ischemic stroke and intracerebral hemorrhage. The most common long-term neurological sequelae are loss of taste/smell, headache, and vertigo. However, there is additional evidence for cognitive impairment among those with severe COVID-19, with 33% of patients discharged from one intensive care unit (ICU) exhibiting clinically relevant inattention, disorientation, and poorly organized movements. Another study utilizing a three-week telephone cognitive screening four weeks after discharge showed that 42% of those who experienced delirium during ICU stay had lasting lower cognitive scores compared to those who did not experience delirium.

The majority of currently available knowledge about neurocognitive symptoms associated with COVID-19 comes from cross-sectional studies of patients in the acute setting. Existing data suggests that following hospitalization, COVID-19 survivors may most frequently demonstrate deficits in letter-cued verbal fluency and executive function. However, this body of research is in its early stages and further investigation is needed. The model of traditional face-to-face cognitive testing using paper and pencil instruments is poorly suited to a global infectious disease pandemic. The Defense Automated Neurobehavioral Assessment (DANA) is a battery of cognitive tests delivered via an electronic tablet or smartphone. The platform allows higher temporal precision and frequency of measurement than traditional neuropsychological methods while including previously standardized cognitive tests and allowing individuals to repeatedly self-administer the battery in the individuals' own homes without examiner supervision. Hence, the DANA battery bypasses several of the major limitations associated with in-person cognitive exams.

ELIGIBILITY:
Inclusion Criteria:

* Have documented pulmonary illness treated in the PACT clinic.
* Have access to an internet-connected electronic device (e.g., Android or iOS phone or tablet) able to perform DANA.
* Agree to participate in seven DANA assessments.
* Be proficient in use of the English language.
* Willing and able to consent to the study.

Exclusion Criteria:

* During the testing phase, plans to undergo treatment with documented lasting neurocognitive effects that will confound DANA assessments, including but not limited to: neurosurgery, chemotherapy, radiation therapy, electroconvulsive therapy, and cardiac surgery.
* During the testing phase, sustains injury or disease state unrelated to reason for PACT admission with documented lasting neurocognitive effects that will confound DANA assessments, including but not limited to: traumatic brain injury (as determined by study clinician).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants must have a documented pulmonary illness due to COVID and being treated in the PACT clinic. They should have access to an internet-connected electronic device (e.g., Android or iOS phone or tablet) able to use the DANA app.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Cognitive dysfunction trajectory | upto 6 months
  ● Characterize the nature (i.e., pattern of cognitive deficits) and trajectory of cognitive dysfunction among those treated for COVID-19 with high temporal resolution repeatedly for up to 6 months using the DANA.

SECONDARY OUTCOMES:
DANA validation | upto 6 months
  ● Validate DANA results against traditional neuropsychological test results collected as part of routine clinical care.

CONTACTS AND LOCATIONS:
Overall Officials: Anupama Kumar, MBBS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Psychiatry department, Baltimore, Maryland, United States